CLINICAL TRIAL: NCT01951001
Title: Fixed-dose vs. Phenotype-based PrAsugrel Dose to MATCH Therapeutic Zone in Asians With Acute Coronary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gyeongsang National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-MATCH; 2013-05-002-004 (Other: GNUH IRB)
Record Dates: First submitted 2013-09-23; First posted 2013-09-26 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-07

CONDITIONS: Acute Coronary Syndrome; Platelet Thrombus; Bleeding
Keywords: Acute Coronary Syndrome, Asians, platelet, prasugrel
MeSH Terms: conditions — Acute Coronary Syndrome; Hemorrhage | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group 1 (Active Comparator): Fixed-dose Prasugrel of 10 mg/d
  Interventions: Drug: Prasugrel
- group 2 (Active Comparator): Fixed-dose Prasugrel of 5 mg/d
  Interventions: Drug: Prasugrel
- group 3 (Active Comparator): Phenotype-based prasugrel dose
  * If patients show PRU < 85, prasugrel dose will be reduced by 5 mg/d.
  * If patients show PRU ≥ 85, prasugrel dose will continue 10 mg/d.
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Prasugrel — For fixed-dose group, patients will receive prasugrel 10 or 5 mg/d for 1 month Irrespective of platelet function test.

SUMMARY:
The purpose of this study is to determine whether the fixed-dose (prasugrel 10 mg/d vs. 5 mg/d) vs. phenotype (platlet function test by VerifyNow P2Y12 assay)-based prasugrel dose adjustment can match therapeutic zone of platelet reactivity in PCI-treated Asians with acute coronary syndrome

DETAILED DESCRIPTION:
The combination of clopidogrel and aspirin has been the mainstay treatment strategy to prevent ischemic events in a wide spectrum of patients with high-risk coronary artery disease. Multiple lines of evidence have demonstrated that patients who are poor responders or who have high on-clopidogrel platelet reactivity (HPR) to adenosine diphosphate (ADP) are at increased risk of post-percutaneous coronary intervention (PCI) ischemic event occurrence. A consensus paper suggested the cutoffs of HPR determined by various platelet function tests to be used for personalized antiplatelet therapy. In addition, several clinical studies have reported that patients with low on-treatment platelet reactivity (LPR) can be related with increased risk of serious bleeding following PCI.

Although multiple coronary risk factors can influence the response to clopidogrel, the cytochrome P450 (CYP) 2C19 loss-of-function allele is a major component in determining the level of platelet reactivity and the prevalence of HPR during clopidogrel treatment. There are multiple CYP2C19 alleles associated with loss-of-function (*2-*8), and interethnic differences in loss-of-function allele carriage exist (Table 1).4 Approximately 30% of Caucasians are the CYP2C19 loss-of-function allele carriers with vast majority carry the *2 allele. However, ~ 65% of East Asians carry the CYP2C19 loss-of-function allele; ~50% carry the *2 allele and the rest carry the *3 allele. Furthermore, the influence of the CYP2C19*3 allele on the antiplatelet response to clopidogrel seems greater compared with the CYP2C19*2 allele.6 It has been suggested that the high prevalence of CYP2C19 loss-of-function allele carriage in East Asians may explain the higher prevalence of HPR during clopidogrel treatment (at least 40% during standard-dose administration).

However, despite the higher prevalence of HPR, numerous prospective clinical studies and registry data have shown that East Asians have similar or even lower rates of post-PCI ischemic event occurrence during clopidogrel therapy compared with Caucasians- the "East Asian paradox". Intriguingly, studies in PCI-treated East Asians have reported higher HPR cutoffs compared with HPR cutoffs obtained from the Western population (252.5-288 vs. 208-235 P2Y12 reaction units [PRU] by the VerifyNow P2Y12 assay). The level and relative contribution of HPR to post-stenting ischemic event occurrence in East Asians may differ from the Western population.

Even though East Asians have shown the low level of platelet inhibition during clopidogrel treatment, accompanying risk of post-PCI serious bleeding in East Asians was highest compared with other races in the CHSRISMA (Clopidogrel for High Atherothrombotic Risk and Ischemic Stabilization, Management, and Avoidance) study.16 Moreover, the suggested cutoff of LPR in PCI-treated Koreans appeared higher compared with that in Caucasians (e.g. VASP-P index 30% vs. 17%). Taken together, East Asians may have an intrinsically reduced risk of arterial thrombosis leading to an increased therapeutic zone of platelet reactivity to ADP compared with Caucasians (the increased cutoffs of LPR and HPR).

# Are there ethnic differences in thrombogenecity? Arterial thrombosis is platelet rich and superimposed on ruptured and inflamed atherosclerotic lesions.18 However, experimental studies suggest that arterial and venous thrombosis are finely regulated processes involving a highly complex interplay between platelets and other blood cells, soluble plasma proteins, and the vessel wall.18,19 The convincing associations of arterial thrombosis to coagulation system and inflammation have been repeatedly demonstrated in multiple clinical trials: fibrinogen, factor V Leiden (G1691A) and prothrombin G20210A gene mutations, high-sensitivity C-reactive protein (CRP) and so on.

To date, there is no definite evidence to suggest that differences in intrinsic platelet function exist between races. However, there are numerous data suggesting inter-ethnic differences in coagulation, fibrinolytic activity, and inflammation. Several population-based clinical trials have reported different incidences of venous thromboembolism (VTE) across races.23,24 In most studies, patients of Asian descent appear to have a lower rate of VTE than other races. Prevalence of arterial thrombosis also has been shown to increase in black race compared with non-black race. This disparity between the races has been partially explained by genetic risk factors.24 In the Multi-ethnic Study of Atherosclerosis (MESA) study evaluating multiple hemostatic factors and plasma endothelial activation markers in individuals living in the USA, African Americans generally had the most thrombogenic and dysfunctional endothelial profile, followed by Hispanics and Caucasians with similar levels, and finally East Asians. A growing body of evidence has demonstrated different levels of inflammation between the races, in which East Asians appear to have the lowest level of inflammation.

In summary, East Asians appear to have a less prothrombotic state compared with African Americans and Caucasians. The latter observation may explain why the East Asian population has a lower risk of ischemic event occurrence and a higher propensity for bleeding during clopidogrel treatment after PCI.

# Future direction of "ethnicity/phenotype-based antiplatelet therapy" Two large-scale, prospective clinical trials (Trial to Assess Improvement in Therapeutic Outcomes by Optimizing Platelet Inhibition With Prasugrel-TIMI 38 [TRITON-TIMI 38] and PLATelet Inhibition and Patient Outcomes [PLATO])30,31 evaluating the clinical efficacy and safety of potent P2Y12 receptor inhibitors (prasugrel and ticagrelor) in ACS patients demonstrated the superiority of strong platelet inhibition to prevent the occurrence of ischemic events compared with clopidogrel treatment. However, the recent "real world" clinical data from Western population have shown that ACS patients with LPR (about 30% of total cohort) have the increased risk of serious bleeding (e.g. 15.5% of TIMI minor plus major bleeding during 1-year prasugrel treatment). In the era of potent P2Y12 receptor inhibitors, the concept of LPR and overcoming the risk of bleeding may be the emerging target in the field of platelet research.

Because PLATO and TRITON TIMI-38 enrolled a limited number of Asians (~3% of total cohort), it is difficult to draw reliable conclusions regarding whether these potent P2Y12 receptor inhibitors will provide similar benefits in East Asians compared with other races. Aforementioned, East Asians may have an intrinsically reduced risk of arterial thrombosis leading to an increased therapeutic zone of platelet reactivity compared with Caucasians. Like most cardiovascular drugs, marked interethnic differences in pharmacokinetics and pharmacodynamics of prasugrel exist. Exposure of the active metabolite and platelet inhibition during prasugrel treatment was higher in East Asians including Chinese, Japanese, and Korean populations compared with Caucasians even after adjustment for body weight. In a recent pharmacodynamic study including stented Koreans, a 10 mg/d of prasugrel achieved the lowest level of PRU compared with 5 mg/d of prasugrel and 75 mg/d of clopidogrel (80.1 ± 45.9 vs.163.1 ± 61.2 vs. 214.0 ± 69.1, p < 0.001). About two thirds of 10 mg/d prasugrel group met the criteria of LPR (≤ 94 PRU), which can support that 10 mg/d of prasugrel is so strong to increase the risk of serious bleeding in most of East Asians.

Taken together, the optimal dosage of antiplatelet regimens and the inhibitory level of the target pathway may differ between the races. In East Asians with less thrombogenicity, excessive inhibition of platelet function by potent P2Y12 receptor inhibitors may markedly increase the risk of serious bleeding without protection against post-PCI ischemic event occurrence. Therefore, dedicated investigations in East Asians are required before we can apply Western recommendations for novel antiplatelet therapy in the former population. It is a time to consider the paradigm shift from "one size fits all" to "ethnicity/phenotype-based antiplatelet therapy". We designed the A-MATCH study to cover this unmet need to guarantee clinical efficacy and safety in East Asians with less thrombogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome (unstable angina, NSTEMI, and STEMI)
* Significant coronary artery stenosis (>50% by visual estimate) eligible for coronary stenting
* Between 20 and 75 years of age
* Body weight ≥ 60kg
* Aspirin dose of 100 mg is recommended
* Ability to understand and to comply with the study protocol

Exclusion Criteria:

* Prior history of ischemic or hemorrhagic stroke or transient ischemic attack, or sub-arachnoids hemorrhage
* fibrinolytic or abciximab therapy within 48 hours of entry or randomization into the study
* vitamin K antagonist
* History of intolerance or allergy to ASA or approved thienopyridines (ticlopidine, clopidogrel, or prasugrel)
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* active pathological bleeding or history of bleeding diathesis
* Thrombocytopenia (platelets < 100,000/mm3)
* Severe hepatic impairment (Child Pugh class C).
* a condition associated with poor treatment compliance, including dementia or mental illness

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Proportion matching to the optimal therapeutic zone | 1 month
  "Therapeutic zone" has been defined based on the previous clinical trials (85 ≤ VerifyNow P2Y12 Reaction Unit ≤ 208)

SECONDARY OUTCOMES:
Prevalence of BARC bleeding | 1 month
  BARC Definition for bleeding: defined as type 1, 2, 3 (3a, 3b and 3c), and 5 (5a and 5b), according to the Bleeding Academic Research Consortium classification
  * Type 1 (nuisance or superficial bleeding
  * Type 2 (internal bleeding)
  * Type 3a (TIMI minor bleeding)
  * Type 3b (TIMI major bleeding)
  * Type 3c (life threatening bleeding)
  * Type 4 (CABG-related bleeding)
  * Type 5a (probable fatal bleeding)
  * Type 5b (definite fatal bleeding)
The cutoff of "LPR" in Asians | 1 month
  "LPR" means "low on-treatment platelet reactivity", which can increase the risk of clinically serious bleeding
Proportion matching to Asian therapeutic zone of platelet reactivity | 1 month
  Multiple clinical studies have shown that the cutoff of about 266 PRU is associated with the risk of ischemic event in Asians.
  LPR will be based on the data of the A-MATCh trial.

OTHER OUTCOMES:
Composite of major adverse clinical events (MACE) | 1 month
  MACE includes composite of CV death, non-fatal MI, stent thrombosis, stroke or ischemia-driven TVR

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoon Jeong, MD, PhD, Principal Investigator — Gyeongsang National University Hospital
Locations (1):
- Gyeonsang National University Hospital, Jinju, Gyeonsangnam-do,, South Korea

REFERENCES:
- [Derived] Jeong YH, Oh JH, Yoon HJ, Park Y, Suh J, Lee SW, Lee K, Kim JS, Chun WJ, Park YH, Nam CW, Kim JH, Ahn JH, Hwang SJ, Hwang JY, Tantry US, Gurbel PA, Shin ES. Pharmacodynamic Profile and Prevalence of Bleeding Episode in East Asian Patients with Acute Coronary Syndromes Treated with Prasugrel Standard-Dose versus De-escalation Strategy: A Randomized A-MATCH Trial. Thromb Haemost. 2021 Oct;121(10):1376-1386. doi: 10.1055/a-1346-3300. Epub 2021 Mar 3. PMID 33401330